CLINICAL TRIAL: NCT02228642
Title: A Prospective Investigation Into the Causes, Symptoms, and Outcomes in Patients With Diabetes Who Experience Hypoglycemia During Their Hospitalization
Brief Title: Hypoglycemia in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Mary Korytkowski, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO14030372; PRO14030372 (Other: PRO14030372)
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Diabetes; Hypoglycemia
Keywords: Type 1 diabetes; Type 2 diabetes; Hypoglycemia; Cognition disorders; Inpatient
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with diabetes who develop low blood sugars (hypoglycemia) in the hospital are at risk for losing the ability to develop symptoms that warn them that they are having a low blood sugar. There is almost no available information investigating how the inability to feel symptoms of a low blood sugar contributes to the risk of this happening when people with diabetes are hospitalized. The purpose of this study is to develop a symptom score model that will help to identify patients at risk for low blood sugars in the hospital and to examine what happens to patients who do experience a low blood sugar in the hospital.

DETAILED DESCRIPTION:
Patients who develop recurrent hypoglycemia are predisposed to developing hypoglycemia-associated autonomic failure (HAAF, impaired awareness). There is almost no information investigating the contribution of HAAF as a risk factor for hypoglycemia in hospitalized patients. Our central aim is to develop a validated inpatient hypoglycemic symptom score model to examine HAAF and its correlation with cognitive dysfunction, re-hospitalization rates, inpatient morbidity and mortality.

This will be a prospective non-blinded study performed in a tertiary care center that will include non-critically insulin treated patients with Type 1 and 2 Diabetes. We will identify patients who have experienced moderate hypoglycemia (40-70 mg/dl) or severe hypoglycemia (< 40 mg/dl) within the prior 24 hours by daily generated computerized reports. Participants will be asked to complete a Hypoglycemia Symptom Scores Questionnaire and cognitive testing within 24-36 hours post event. Participants will be contacted at 6 and 12 months following the index hospitalization to obtain information regarding recurrent episodes of hypoglycemia, need for re-hospitalization, and occurrence of any new diabetes related complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes
* Non-critically ill hospitalized surgical and medical patients
* Anticipated length of stay (LOS) >3 days
* Anticipated life expectancy > 1 year
* Mentally competent individuals

Exclusion Criteria:

* Patients who are admitted for hypoglycemia or Diabetic Ketoacidosis
* Anticipated LOS <3 days
* Mentally incompetent individuals defined as any patient with evidence of dementia or delirium recorded in their medical history or progress note
* Patients receiving Total Parenteral Nutrition
* Treatment with high dose narcotic medications
* Patients who would not be able to follow up at 3 to 6 and 9-12 months by telephone call
* Patients with expected life expectancy < 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill hospitalized patients with a diagnosis of diabetes at time of admission using established ADA criteria or prior physician diagnosis who experience a documented episode of hypoglycemia, defined as a blood glucose < 70 mg/dl.
  .
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2014-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hypoglycemia Associated Autonomic Failure in the inpatient setting as assessed by hypoglycemia symptom scores | Within 24-36 hours following a hypoglycemia event.
  Hypoglycemia Symptom Score Questionnaires will be administered to participants in time frame described. These questionnaires include a list of potential autonomic and neuroglycopenic symptoms that can occur in response to hypoglycemia.

SECONDARY OUTCOMES:
Measures of cognitive function following a hypoglycemic event | Within 24 to 36 hours of a hypoglycemia event.
  Cognitive function testing will be performed using the St Louis University Mental Status Exam Survey (SLUMS)

OTHER OUTCOMES:
Adverse events following a hypoglycemic event. | Up to one year following the hypoglycemia event
  Information regarding falls, myocardial infarction, arrhythmia, seizures or other adverse events that occur following the hypoglycemia event will be collected.
Measure of cognitive function | Within 24 to 36 hours of the index hypoglycemic event
  STROOP color word interference test

CONTACTS AND LOCATIONS:
Overall Officials: Mary T Korytkowski, MD, Principal Investigator — University of Pittsburgh School of Medicine, Department of Medicine
Locations (1):
- University of Pittsburgh Medical Center PUH SSY, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided